CLINICAL TRIAL: NCT00150553
Title: A Phase IIIb, Randomized, Double-Blind, Parallel Group Study in Bipolar I Patients to Assess the Efficacy and Safety of SPD417 Administered Once Daily vs Twice Daily in the Treatment of Manic Symptoms
Brief Title: Efficacy and Safety of SPD417 in Treatment of Manic Symptoms in Adults With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Validus Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD417-306
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2006-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

INTERVENTIONS:
Drug: Extended-release carbamazepine

SUMMARY:
The purpose of this study is to compare the efficacy and safety of SPD417 in treating bipolar manic symptoms, when given once daily in the evening vs. twice daily.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for bipolar I disorder
* Screen YMRS score => 16
* Women of childbearing potential agree to take adequate precautions against contraception

Exclusion Criteria:

* Hospitalization required for treatment of psychiatric symptoms
* Patients who meet DSM-IV for ultra-rapid cycling
* History of serious suicide attempt requiring medical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2005-01; Study Completion 2005-10

PRIMARY OUTCOMES:
Score on Young Mania Rating Scale (YMRS) at 12 weeks

SECONDARY OUTCOMES:
Time to remission
Clinical Global Impressions Scale - Bipolar Version
HAM-D and MADRS scales for depression